CLINICAL TRIAL: NCT00264238
Title: An Open-Label Trial of Memantine to Augment Response in the Treatment of Obsessive-Compulsive Disorder
Brief Title: Memantine Augmentation in Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, John J Barry, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUSPO34313
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine open label (Experimental): All subjects knowingly received (open label) memantine for up to 12 weeks with a target dose of 10 mg twice a day (20mg/d) taken orally.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — pharmacological dosing of memantine as adjunctive therapy for treatment-resistant obsessive-compulsive disorder
  Other Names: Namenda

SUMMARY:
The purpose of this study is to determine whether memantine is safe and effective when used as an augmentation to standard treatment for Obsessive-Compulsive Disorder (OCD).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether memantine (Namenda), in doses up to 20 mg/day, will be effective in treating the OCD of adult patients who have not responded to their OCD medication. Memantine is not FDA approved for OCD, but is approved for the treatment of Alzheimer's Disease. Memantine appears to work by regulating the activity of glutamate, one of the brain's specialized messenger chemicals, which may play a role in OCD. All patients in the study will receive memantine; no one will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* suffering from OCD
* Y-BOCS score of 18 or greater
* taking a therapeutic dose of an anti-OCD medication specified in the protocol

Exclusion Criteria:

* diagnosed with a mental disorder other than OCD
* taking tiagabine or pregabalin
* having had a previous trial of memantine
* receiving therapy for OCD
* substance abuse in the last 6 months
* personality disorders sufficiently severe to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Barry, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aboujaoude E, Barry JJ, Gamel N. Memantine augmentation in treatment-resistant obsessive-compulsive disorder: an open-label trial. J Clin Psychopharmacol. 2009 Feb;29(1):51-5. doi: 10.1097/JCP.0b013e318192e9a4. PMID 19142108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2006 to February 2008, participants recruited from the Stanford School of Medicine Department of Psychiatry and Behavioral Sciences OCD clinic and through online adds. Subjects had to have had failed to respond to at least 12 weeks of treatment at an adequate and stable dose of an serotonin reuptake inhibitor (SRI) (YBOCS of GE 18)
Period: Overall Study
Arm/Group | Memantine Open Label
Started | 15
Completed | 14
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Memantine Open Label
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Yale-Brown Obsessive Compulsive Scale [Mean (Standard Deviation); unit: units on a scale] — The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is designed to rate the severity and type of symptoms in patients with obsessive compulsive disorder. In general, the items depend on the patient's report; however, the final rating is based on the clinical judgement of the interviewer. The Y-BOCS is designed to rate symptom severity, not to establish a diagnosis.The scale consists of 10 items summed to determine the level of symptom severity. The total score ranges from 0 to 40 with higher scores indicating greater symptom severity
  units on a scale | 27.4 (5)
Psychiatric comorbid condition [Number; unit: participants]
  Participants with comorbid condition | 8
  Participants without comorbid condition | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) From Baseline to End of Treatment (12 Weeks)
Description: The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is designed to rate the severity and type of symptoms in patients with obsessive compulsive disorder. In general, the items depend on the patient's report; however, the final rating is based on the clinical judgement of the interviewer. The Y-BOCS is designed to rate symptom severity, not to establish a diagnosis.The scale consists of 10 items summed to determine the level of symptom severity. The total score ranges from 0 to 40 with higher scores indicating greater symptom severity
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Responders: Memantine Open Label: Participants who respond to memantine as adjunctive therapy defined as Y-BOCS decrease of greater than or equal to 25% from baseline and a CGI-I rating of "much" or "very much" improved.
- Non-Responders: Memantine Open Label: Participants who did not respond to memantine as adjunctive therapy
Arm/Group | Responders: Memantine Open Label | Non-Responders: Memantine Open Label
Number analyzed (Participants) | 6 | 8
units on a scale
  At baseline | 23.8 (3.5) | 30 (4.4)
  At end of treatment | 13.0 (4.3) | 28.8 (4.7)

2. Secondary Outcome: Mean Change in Montgomery-Asberg Depression Rating Scale (MADRS) From Baseline to End of Treatment (12 Weeks)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on a scale of 0 (no symptoms) to 6 (extreme symptoms) and items are summed. The overall score ranges from 0 to 60. Higher MADRS score indicates more severe depression.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Responders: Memantine Open Label: Participants who respond to memantine as adjunctive therapy; that is, Y-BOCS decrease of greater than or equal to 25% from baseline and a CGI0I rating of "much" or "very much" improved.
Arm/Group | Responders: Memantine Open Label | Non-Responders: Memantine Open Label
Number analyzed (Participants) | 6 | 8
units on a scale
  Mean at baseline | 11.8 (6.6) | 14.9 (8.4)
  Mean at end of treatment | 5.0 (6.5) | 14.6 (10.5)

ADVERSE EVENTS:
Time Frame: 12 weeks of study medication dosing
Arm/Group | Memantine Open Label
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 7/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine Open Label (N=14)
Nausea (Gastrointestinal disorders) | 3 (3) — Mild to moderate, transient in duration
Headache (Nervous system disorders) | 3 (3) — Mild to moderate, transient in duration
Somnolence (Psychiatric disorders) | 1 (1) — Mild to moderate, transient in duration
Night sweats (General disorders) | 1 (1) — Mild to moderate, transient in duration
Light-headedness (Investigations) | 1 (1) — Mild to moderate, transient in duration
Fatigue (Nervous system disorders) | 1 (1) — Mild to moderate, transient in duration

LIMITATIONS AND CAVEATS:
This study is limited by its open-label design, small size, and the presence of comorbidities and concurrent psychotropic medications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes